CLINICAL TRIAL: NCT03574805
Title: A Dose-Escalating, Single-Blind Study to Assess the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of PRS-060 Administered by Oral Inhalation in Subjects With Mild Asthma
Brief Title: Study of Multiple Doses of PRS-060 Administered by Oral Inhalation in Subjects With Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pieris Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRS-060-PCS_07_18
Record Dates: First submitted 2018-06-11; First posted 2018-07-02 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Asthma
Keywords: Asthma; Anticalin; PRS-060; Pieris; IL-4 receptor alpha; IL-13; IL-4
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRS-060 (Active Comparator): PRS-060 or Placebo
  Interventions: Drug: PRS-060
- Placebo (Placebo Comparator): PRS-060 or Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRS-060 — Study drug
  Arms: PRS-060
Drug: Placebo — Inhalant designed to mimic PRS-060
  Arms: Placebo

SUMMARY:
Study of Multiple Doses of PRS-060 Administered by Oral Inhalation in Subjects with Mild Asthma

DETAILED DESCRIPTION:
PRS-060 is a drug candidate being developed for the treatment of asthma. The main purpose of this study is to investigate the safety, tolerability, and pharmacokinetics of multiple doses of PRS-060 administered by inhalation in subjects with mild asthma.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18 to 35
* Subjects who are non-smokers or ex-smokers who have smoked no more than twice in 3 months prior to screening (determined by urine continine < 500 ng/mL, at Screening visit)
* Males and non-pregnant, non-breastfeeding females
* Males who are sexually active with women of childbearing potential must agree to follow a highly effective method(s) of contraception for the duration of treatment with study drug as well as for an additional 90 days post-treatment completion. Women of childbearing potential who are sexually active with a fertile male must agree to follow instructions for double methods of contraception for the duration of their participation in the trial and for 90 days post-treatment completion
* Documented diagnosis of mild asthma
* 18 to 55 years of age
* Lung function ≥ 70% predicted for FEV1 and FEV1/FVC ratio ≥ 0.7
* FeNO ≥ 35 ppb at Screening and during pre-qualification for the study

Exclusion Criteria:

* History or clinical manifestations of any clinically significant medical disorder that, in the opinion of the investigator, may put the subject at risk because of participation in the study, influence the results of the study, or affect the subject's ability to participate in the study
* A history of drug or alcohol abuse
* History of, or known significant infection including hepatitis A, B, or C, Human immunodeficiency Virus (HIV), tuberculosis (i.e., positive result for interferon [IFN]-γ release assay [IGRA], QuantiFERON® TB-Gold), that may put the subject at risk during participation in the study
* History of cancer within the last 10 years (20 years for breast cancer) except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured. Any history of lymphoma is not allowed
* Any clinically significant illness, infection, medical/surgical procedure, or trauma within 4 weeks of Day 1 or planned inpatient surgery or hospitalization during the study period
* Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the Principal Investigator
* Significant history of recurrent ongoing 'dry eye syndrome' of any cause that may be chronic or acute, that may affect the interpretation of safety data associated with the potential for ADAs targeted to PRS-060 (structurally related to tear lipocalin)
* Subjects who have received live or attenuated vaccine in the 4 weeks prior to Day 1
* Subjects with a disease history suggesting abnormal immune function
* History of anaphylaxis following any biologic therapy and known history of allergy or reaction to any component of the investigational product formulation
* Inability to communicate well with the Investigator (i.e., language problem, poor mental development, or impaired cerebral function)
* Participation in any clinical study for a New Chemical Entity within the previous 16 weeks or a marketed drug clinical study within the previous 12 weeks or within 5 half-lives, whichever is the longer, before the first dose of study drug
* Donation of 450 mL or more blood within the previous 12 weeks
* Women who are pregnant, or breastfeeding, or planning to become pregnant within the study period or 90 days post-treatment completion
* Males who are sexually active with a female partner of childbearing potential and who have not had a vasectomy and who do not agree to a highly effective method of contraception from Day 1 to 90 days post-treatment completion. Females of childbearing potential who are sexually active with a fertile male partner who do not agree to double methods of contraception with at least one barrier from Day 1 to 90 days post-treatment completion
* Life-threatening asthmatic episode in the past
* C-reactive protein (CRP) above 5 mg/L
* Use of the following medicines within the specified time before screening:

  * Long-acting β2 agonists; none for 4 weeks prior to Screening
  * Anti-IgE or anti-IL-5 therapy; for 6 months prior to Screening
  * Inhaled corticosteroids (> 500 μg per day of beclometasone dipropionate [BDP] or equivalent) within 16 weeks prior to Screening
  * Inhaled corticosteroids; none for 4 weeks prior to screening
  * Oral or injectable steroids for the treatment of asthma or respiratory tract infection within 5 years prior to Screening
  * Intranasal steroids within 4 weeks prior to Screening
  * Topical steroids within 4 weeks prior to Screening
  * Leukotriene antagonists within 2 weeks prior to Screening
  * Xanthines (excluding caffeine), anticholinergics, or cromoglycate within 1 week prior to Screening
  * PRS-060 at anytime

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) after an inhaled dose of PRS-060 | From time of dose until 30 days after dosing
  The number of participants with treatment related AEs as assessed by current approved CTCAE version
Change in blood pressure | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess blood pressure (systolic and diastolic) as a criterion of safety and tolerability variables as measured in mm Hg)
Change in heart rate | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in beats per minute (BPM) as a criterion of safety and tolerability variables
Change in body temperature | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in body temperature in degrees Celsius as a criterion of safety and tolerability variables
Change in electrocardiograms (ECGs) | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in cardiovascular system function (change in QTC parameters) as a criterion of safety and tolerability variables
Change in forced expiratory volume 1-second (FEV1) as part of spirometry | Screening, during treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in FEV1 as measured in mL as part of spirometry
Change in forced vital capacity (FVC) as part of spirometry | Screening, during treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in FVC as measured by mL
Change in peak expiratory flow rate (PEFR) as part of spirometry | Screening, during treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in PEFR as measured in L/min
Change in sodium levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To asses changes in sodium levels as measured in mmol/L
Change in potassium levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in potassium levels as measured in mmol/L
Change in chloride levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days)
  To assess changes in chloride levels as measured in mmol/L
Change in bicarbonate levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in bicarbonate levels as measured in mmol/L
Change in blood urea nitrogen (BUN)/Urea levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes BUN/Urea levels as measured in mmol/L
Change in creatinine levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in creatinine levels as measured in umol/L
Change in total protein levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in total protein levels as measured in g/L
Change in albumin levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in albumin levels as measure in g/L
Change in alkaline phosphate (ALP) levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in ALP levels as measured in U/L
Change in ALT levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in ALT levels as measured in U/L
Changes in AST levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in AST levels as measured in U/L
Change in total bilirubin levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in total bilirubin levels as measured in umol/L
Change in direct bilirubin levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in direct bilirubin levels as measured in umol/L
Change in indirect bilirubin levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in indirect bilirubin levels as measured in umol/L
Change in amylase levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in amylase levels as measured in U/L
Change in lipase levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in lipase levels as measured in U/L
Change in uric acid levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in uric acid levels as measured in mmol/L
Change in creatine kinase (CK) levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in CK levels as measured in U/L
Change in calcium levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in calcium levels as measured in mmol/L
Change in magnesium levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in magnesium levels as measured in mmol/L
Change in lactate dehydrogenase (LDH) levels as part of standard serum chemistry panel. | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in LDH levels as measure in U/L
Change in total immunoglobulin (IgG) levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in total IgG levels as measured in g/L
Changes in total immunoglobulin (IgA) levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in total IgA levels as measured in g/L
Changes in total immunoglobulin (IgE) levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in total IgE levels as measured in lU/mL
Change in total immunoglobulin (IgM) levels as part of standard serum chemistry panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in total IgM levels as measured in g/L
Change in hematocrit as part of standard hematology panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in total hamatocrit levels as measured by %
Change in hemoglobin levels as part of standard hematology panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in hemoglobin levels as measured by g/L
Change in red blood cells (RBC) counts as part of standard hematology panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in red blood cells (RBC) counts as measured by 10^12/uL
Change in platelet (PLT) counts as part of standard hematology panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in PLT counts as measured by 10^9/uL
Change in white blood cells (WBC) counts as part of standard hematology panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in white blood cell (WBC) counts as measured by 10^9/uL
Change in neutrophil percentage as part of standard hematology panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in neutrophil percentages as measured by %
Change in lymphocyte percentage as part of standard hematology panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in lymphocyte percentage as measured by %
Change in eosinophil percentage a part of standard hematology panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in eosinophil percentage as measured by %
Change in basophil percentage as part of standard hematology panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes basophil percentages as measured by %
Change in monocyte percentage as part of standard hematology panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in monocyte percentage as measured by %
Change in clarity as part of a standard urinalysis panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in clarity of the urine sample
Change in specific gravity as part of a standard urinalysis panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in specific gravity of the urine sample
Change in pH as part of a standard urinalysis panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in pH of the urine sample
Change in protein levels as part of a standard urinalysis panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in protein levels of the urine sample
Change in glucose levels as part of a standard urinalysis panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in glucose levels of the urine sample as measured by a positive or negative result.
Change in ketone levels as part of a standard urinalysis panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in ketone levels of the urine sample as measured by a positive or negative result
Change in blood levels as part of a standard urinalysis panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in blood levels of the urine sample as measured by a positive or negative result.
Change in nitrite levels as part of a standard urinalysis panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in nitrite levels of the urine sample
Change in leukocyte esterase levels as part of a standard urinalysis panel | Screening, during treatment, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  To assess changes in leukocyte esterase levels of the urine sample

SECONDARY OUTCOMES:
PK assessment: Cmax (observed maximum serum concentration taken directly from the individual concentration-time curve) | During treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  Evaluation of the PK after receiving PRS-060
PK assessment: Tmax (time to reach maximum serum concentration, taken directly from the individual concentration-time curve) | During treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  Evaluation of the PK after receiving PRS-060
PK assessment: t1/2(terminal half-life) | During treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  Evaluation of the PK after receiving PRS-060
PK assessment: AUC (0-last) (area under the serum concentration-curve from time zero to the time of last quantifiable analyte concentration) | During treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  Evaluation of the PK after receiving PRS-060
PK assessment: AUC (area under the concentration-time curve in the serum zero [pre-dose] extrapolated to infinite time) | During treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  Evaluation of the PK after receiving PRS-060
PK assessment: AUC (0-24) (area under the plasma concentration-curve) | During treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  Evaluation of the PK after receiving PRS-060
PK assessment: Vz/F (apparent volume of distribution during terminal phase) | During treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  Evaluation of the PK after receiving PRS-060
PK assessment: CL/F (apparent oral clearance estimated as dose divided by AUC) | During treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  Evaluation of the PK after receiving PRS-060
PK assessment of urine | During treatment and confinement
  Evaluation of PRS-060 levels in the urine after receiving PRS-060
Serum ADA assessment using bridging Immunoassay Enhanced Chemiluminescence (ECL) method | During treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  Evaluation of potential development of ADAs against PRS-060
FeNO assessment | Screening, during treatment and confinement, 7 days after dosing (±1 day), and 30 days after dosing (±3 days).
  Evaluation of FeNO after receiving PRS-060 or placebo

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Q-Pharm, Herston, Queensland
  - CMAX, Adelaide, South Australia
  - Nucleus Network Limited, Melbourne, Victoria
  - Linear, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided